CLINICAL TRIAL: NCT04354818
Title: Coronavirus Outcomes Registries in Immunocompromised Individuals Australia (CORIA): a Multisite Registry and Optional Biorepository in People With COVID-19 and Selected Conditions Affecting Immune Function
Brief Title: Coronavirus (COVID-19) Outcomes Registries in Immunocompromised Individuals Australia (CORIA)
Acronym: CORIA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kirby Institute (Other Government)
Collaborators: St Vincent's Hospital, Sydney (Other); Garvan Institute of Medical Research (Other); Westmead Hospital, Sydney, Australia (Unknown); Blacktown Hospital, Sydney, Australia (Unknown); Holdsworth House Medical Practice (Other); Royal North Shore Hospital (Other); Melanoma Institute Australia (Other); Prince of Wales Hospital, Sydney (Other Government); Gilead Sciences (Industry); Cancer Institute NSW (Unknown); Cancer Council New South Wales (Other); Positive Life NSW (Unknown); St George Hospital, Australia (Other); Liverpool Hospital, Sydney (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-04-CORIA
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: HIV-1-infection; Cancer; Primary Immune Deficiency Disorder; Immunosuppression Disorders; COVID-19
MeSH Terms: conditions — Neoplasms; Primary Immunodeficiency Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- People living with HIV
- Recipients of Solid Organ Transplants
- People Living with Cancer
- People with acquired immunodeficiency: Patients with acquired immunodeficiency associated with other immunosuppressive therapy.
- People with primary immunodeficiency

SUMMARY:
CORIA is an observational cohort study of immunosuppressed populations who test positive for COVID-19. This includes people living with HIV, cancer, acquired immunodeficiency associated with other immunosuppressive therapy, primary immunodeficiency and recipients of a solid organ transplant. Participants will have routine clinical data collected with optional baseline collection and storage of a blood sample for storage . The study will be conducted in up to 30 sites within Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting (in person or via telemedicine) for evaluation because they:

   * Have clinical symptoms consistent with for COVID-19:
   * Fever (≥ 37.8 °C) on examination OR patient reported fever (≥ 37.8 °C) or feverishness (felt febrile but did not take temperature) OR any of, cough, sore throat, shortness of breath, rhinorrhoea, headache, chills, generalise myalgia, malaise, fatigue, confusion, diarrhea, nausea or vomiting
   * Have been contacted because they have been identified as a contact to a confirmed case
   * Have been contacted and told they tested positive for COVID-19
2. Have one of the following conditions affecting immune function:

   * Known or suspected primary immunodeficiency, defined as a predisposition to infection associated with an apparent or presumed deficit of immune function
   * On immunosuppressive therapy
   * Treatment with immune checkpoint inhibitors within 36 months of enrolment date
   * HIV infection
   * Diagnosis of cancer within 36 months of enrolment date, excluding superficial basal cell and squamous cell carcinomas
   * Solid organ transplantation
3. For optional biobanking only, ability to provide informed consent

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 years or older with a known condition affecting immune function (Primary Immune Deficiency, on Immunosuppressive Therapy, on Immune checkpoint inhibitors within 36 months of study enrolment, HIV infection, recipient of Solid Organ Transplant or diagnosis of Cancer within 36 months of study enrolment, excluding superficial basal cell and squamous cell carcinomas) presenting with clinical symptoms consistent with COVID-19 or a known contact to a confirmed case or known to be COVID-19 positive.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-04-27 (Estimated); Study Completion 2022-04-27 (Estimated)

PRIMARY OUTCOMES:
percentage of patients who required hospitalisation, developed severe illness (ICU admission) or died | Day 28

SECONDARY OUTCOMES:
percentage of patients who required hospitalisation, developed severe illness (ICU admission) or died | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Polizzotto, MD, Principal Investigator — Kirby Institute
Locations (11):
- Australia (11):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - East Sydney Doctors, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Concord Hospital, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Melanoma Institute Australia, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No